CLINICAL TRIAL: NCT01227577
Title: A Single-arm, Open-label, Multi-center Study of Complete Molecular Response (CMR) in Adult Patients With Newly Diagnosed Philadelphia Chromosome Positive (Ph+) Chronic Myelogenous Leukemia in Chronic Phase (CML-CP)
Brief Title: CMR Rate of Newly Diagnosed CML-CP Patients Treated With Nilotinib
Acronym: MACS1428
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CAMN107AUS28
Record Dates: First submitted 2010-10-21; First posted 2010-10-25 (Estimated); Results first posted 2016-02-08 (Estimated); Last update posted 2016-02-08 (Estimated); Status verified 2016-01

CONDITIONS: Chronic Myelogenous Leukemia in Chronic Phase
Keywords: CML; Chronic Myelogenous Leukemia; Leukemia; CML-CP; Nilotinib
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Leukemia | interventions — nilotinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Nilotinib (Experimental): Participants received 300 mg twice daily (b.i.d.). Dose increases to 400 b.i.d. were permitted, per Investigator's discretion.
  Interventions: Drug: Nilotinib

INTERVENTIONS:
Drug: Nilotinib — Nilotinib was supplied as 150 mg and 200 mg hard gelatin capsules.

SUMMARY:
"This is a single-arm, open-label, multi-center study of complete molecular response (CMR) in adult patients with newly diagnosed Philadelphia chromosome positive (Ph+) chronic myelogenous leukemia in chronic phase (CML-CP). The study is designed to evaluate early and deep molecular responses up to 4 years on nilotinib treatment. The primary end point is Rate of confirmed CMR in newly diagnosed Philadelphia chromosome positive CML-CP patients."

ELIGIBILITY:
Inclusion Criteria:

Patients with Ph+ CML-CP within 3 months of diagnosis. Male or female patients' ≥ 18 years of age. Patients must have adequate end organ function.

Exclusion Criteria:

Previously documented T315I mutation. Other CML treatment is an exclusion criteria with the following exception: While awaiting study start, patients may be treated with anagrelide (no treatment duration limit), hydroxyurea (no treatment duration limit), and/or up to a 14 day supply of a tyrosine kinase inhibitor (TKI) approved by the FDA for frontline treatment. Patients taking a TKI prior to study entry must have at least a one day washout from their last dose of medication and have recovered from any side effects of such therapy.

Impaired cardiac function as defined by the protocol. Patients with contraindications to receiving nilotinib, including concomitant medications.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Actual)
Dates: Start 2010-11; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (32):
- United States (32):
  - Pacific Cancer Medical Center, Inc., Anaheim, California
  - Providence St. Joseph Medical Center Roy&Patricia Disney Fam Cancer, Burbank, California
  - Bay Area Cancer Research Dept.ofBayAreaCancerResearch, Concord, California
  - St. Jude Heritage Medical Group Virginia Crosson Cancer Center, Yorba Linda, California
  - Sarah Cannon Research Institute SCRI, Jacksonville, Florida
  - Advanced Medical Specialties, Miami, Florida
  - Pasco Hernando Oncology, New Port Richey, Florida
  - Georgia Regents University MedCollege of GA Cancer Ctr 2, Augusta, Georgia
  - Stroger Cook County Hospital Division of Hematology & Onc, Chicago, Illinois
  - Louis A. Weiss Memorial Hospital, Chicago, Illinois
  - Indiana Blood and Marrow Institute, Beach Grove, Indiana
  - Cancer Center of Kansas, Witchita, Kansas
  - LSU HEALTH SCIENCES CENTER/ LSU SCHOOL OF MEDICINE Feist-Weiller Cancer Center(3), New Orleans, Louisiana
  - University of Maryland, Baltimore, Maryland
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Henry Ford Hospital, Detroit, Michigan
  - St. Louis University Cancer Center, St Louis, Missouri
  - University of Nebraska Medical Center University of Nebraska Med Ctr, Omaha, Nebraska
  - Hackensack University Medical Center Dept.of HackensackUniv.MedCtr., Hackensack, New Jersey
  - University of Rochester Medical Ct James P Wilmot Cancer Ctr, Rochester, New York
  - Montefiore Medical Center, The Bronx, New York
  - Duke University Medical Center Duke University Med Ctr, Durham, North Carolina
  - Oregon Health & Science University, Portland, Oregon
  - Cancer Centers of the Carolinas Cancer Center, Greenville, South Carolina
  - Chattanooga Oncology and Hematology Assoicates, PC Chattanooga Oncology, Chattanooga, Tennessee
  - The Jones Clinic, Germantown, Tennessee
  - Tennessee Oncology Sarah Cannon Research Inst., Nashville, Tennessee
  - Baylor Research Institute Baylor Research Institute (17), Dallas, Texas
  - Oncology Consultants Oncology Consultants, P.A., Houston, Texas
  - Millennium Oncology, Houston, Texas
  - University of Virginia, Charlottesville, Virginia
  - Providence Regional Cancer Partnership, Everett, Washington

REFERENCES:
- [Derived] Berdeja JG, Heinrich MC, Dakhil SR, Goldberg SL, Wadleigh M, Kuriakose P, Cortes J, Radich J, Helton B, Rizzieri D, Paley C, Dautaj I, Mauro MJ. Rates of deep molecular response by digital and conventional PCR with frontline nilotinib in newly diagnosed chronic myeloid leukemia: a landmark analysis. Leuk Lymphoma. 2019 Oct;60(10):2384-2393. doi: 10.1080/10428194.2019.1590569. Epub 2019 Mar 26. PMID 30912699

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Nilotinib
Started | 128
Completed | 93
Not Completed | 35
Not completed — Protocol deviation | 3
Not completed — Death | 3
Not completed — Administrative problems | 2
Not completed — Lost to Follow-up | 1
Not completed — Withdrawal by Subject | 4
Not completed — Lack of Efficacy | 5
Not completed — Adverse Event | 17

BASELINE CHARACTERISTICS:
Arm/Group | Nilotinib
Number analyzed (Participants) | 128
Age, Continuous [Mean (Standard Deviation); unit: Years] | 55.6 (14.99)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 64
  Male | 64

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Confirmed Complete Molecular Response (CMR)
Description: CMR was defined as at least 4.5 log reduction of breakpoint cluster region gene/Abelson proto-oncogene (Bcr-Abl) transcipts from the standardized baseline on the international scale (equivalent to Bcr-Abl <=0.0032% IS) with a minimum of 25,614 ABL control copies. CMR was to be confirmed by a second polymerase chain reaction (PCR) sample drawn 3 months later where the results should be less than or equal to 0.0032% with a minimum of 25,614 Abelson proto-oncogene (ABL) control copies.
Time Frame: 4 years
Population: Full Analysis Set (FAS): The FAS included all randomized participants who received at least one dose of study drug.
Measure: Number; unit: Participants
Arm/Group | Nilotinib
Number analyzed (Participants) | 128
Participants | 34

2. Secondary Outcome: Number of Participants With Complete Cytogenetic Response (CCyR) and Major Molecular Response (MMR)
Description: CCyR was defined as 0% Philadelphia chromosome-positive (Ph+) metaphases in the bone marrow. MMR was defined as a 3 log reduction of Bcr-Abl transcripts from the standardized baseline on the international scale (equivalent to Bcr-Abl ≤ 0.1% IS).
  Bcr-Abl transcripts assessed by peripheral blood quatitative real time polymerase chain reaction (RQ-PCR) were used for the determination of all molecular responses.
Time Frame: 4 years
Population: Full Analysis Set (FAS): The FAS included all randomized participants who received at least one dose of study drug.
Measure: Number; unit: Participants
Arm/Group | Nilotinib
Number analyzed (Participants) | 128
Participants
  CCyR | 93
  MMR | 94

3. Secondary Outcome: Time to CMR, CCyR and MMR
Description: Time to CMR, CCyR, and MMR was defined as the time from the date of enrollment to the date of first documented CMR, CCyR and MMR, respectively.
Time Frame: 4 years
Population: Of the 128 participants analyzed, 34 participants achieved CMR within 18 months of treatment, 93 participants achieved CCyR and did not experience loss of CCyR during the study, and 94 participants achieved MMR with up to 24 months of treatment (most achieved MMR within 12 months of treatment).
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Nilotinib
Number analyzed (Participants) | 128
Months
  CMR (n=34) | NA [NA to NA] — The median could not be calculated due to insufficient events.
  CCyR (n=93) | 5.5 [4.07 to 5.55]
  MMR (n=94) | 5.7 [5.55 to 7.66]

4. Secondary Outcome: Duration of CMR, CCyR and MMR
Description: Duration of CMR, CCyR and MMR were defined as the time from the first date of achievement of the response to the date of first documented loss of the response.
Time Frame: 4 years
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Months
Arm/Group | Nilotinib
Number analyzed (Participants) | 128
Months
  CMR (n=34) | 7.97 (3.705)
  CCyR (n=93) | NA (NA) — None of the participants experienced loss of CCyR during the study.
  MMR (n=94) | 4.86 (5.003)

5. Secondary Outcome: Number of Participants With Progression to Accelerated Phase/Blastic Crisis (AP/BC)
Description: Progression to AP/BC is defined as loss of CCyR, MMR, and CMR and was summarized by frequencies and percentages.
Time Frame: 4 years
Population: Full Analysis Set (FAS): The FAS included all randomized participants who received at least one dose of study drug.
Measure: Number; unit: Participants
Arm/Group | Nilotinib
Number analyzed (Participants) | 128
Participants | 1

6. Secondary Outcome: Time to Progression of AP/BC
Description: Time to progression of AP/BC was defined as the time from the date of the first dose of study drug to the date of first documented progression of AP/BC.
Time Frame: 4 years
Population: Of the 128 participants analyzed, 1 participant experienced progression to AP/BC.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Nilotinib
Number analyzed (Participants) | 128
Months | NA [NA to NA] — The median could not be calculated due to an insufficient number of events.

7. Secondary Outcome: Number of Participants With Loss of CCyR, MMR and CMR
Description: Rate of loss of CMR was defined as an increase in the Bcr-Abl transcripts to greater than 0.0032% IS. Rate of loss of CCyR was defined as an increase in the Ph+ bone marrow cells to greater than 0%. Rate of loss of MMR was defined as an increase in the Bcr-Abl transcripts to greater than 0.1% IS.
Time Frame: 4 years
Population: Numbers are based on the total number of participants who achieved and experienced loss of CMR (34 participants), CCyr (93 participants) and MMR (94 participants), respectively.
Measure: Number; unit: Participants
Arm/Group | Nilotinib
Number analyzed (Participants) | 128
Participants
  CMR (n=34) | 6
  CCyR (n=93) | 0
  MMR (n=94) | 13

8. Secondary Outcome: Number of Participants With CMR Who Were Dosed to 400 mg b.i.d.
Description: as for outcome 1
Time Frame: 4 years
Population: Of the 128 participants analyzed, 3 participants received an escalated dose of 400 mg b.i.d.
Measure: Number; unit: Participants
Arm/Group | Nilotinib
Number analyzed (Participants) | 3
Participants | 0

9. Secondary Outcome: Event-free Survival, Progression-free Survival and Overall Survival
Description: Event-free survival was defined as the time from the date of enrollment to the date of first occurrence of any of the following: loss of Complete Hematological Response (CHR), loss of CCyR, loss of Partial Cytogenetic Response (PCyR), progression to the accelerated phase or blast crisis, and death from any cause. Progression-free survival was defined as the time from the date of enrollment to the date of first occurrence of any of the following: progression to the accelerated phase or blast crisis, death, and loss of CMR. Overall survival was defined as the time from the date of enrollment until death due to any cause.
Time Frame: 4 years
Population: Full Analysis Set (FAS): The FAS included all randomized participants who received at least one dose of study drug.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Nilotinib
Number analyzed (Participants) | 128
Months
  Event-free | NA [NA to NA] — Median could not be calculated due to an insuffient number of events.
  Progression-free | NA [NA to NA] — Median could not be calculated due to an insuffient number of events.
  Overall | NA [NA to NA] — Median could not be calculated due to an insuffient number of events.

ADVERSE EVENTS:
Arm/Group | Nilotinib
Serious Adverse Events (participants affected / at risk) | 27/128
Other Adverse Events (participants affected / at risk) | 122/128
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Nilotinib (N=128)
Neutropenia (Blood and lymphatic system disorders) | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 2
Atrial fibrillation (Cardiac disorders) | 1
Myocardial infarction (Cardiac disorders) | 3
Palpitations (Cardiac disorders) | 1
Hyperthyroidism (Endocrine disorders) | 1
Toxic nodular goitre (Endocrine disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 4
Gastritis (Gastrointestinal disorders) | 1
Intestinal obstruction (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Oesophagitis (Gastrointestinal disorders) | 1
Pancreatitis (Gastrointestinal disorders) | 3
Small intestinal obstruction (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Chest pain (General disorders) | 2
Pyrexia (General disorders) | 1
Cholecystitis acute (Hepatobiliary disorders) | 1
Device related infection (Infections and infestations) | 1
Gastroenteritis (Infections and infestations) | 1
Gastroenteritis viral (Infections and infestations) | 1
Pharyngitis streptococcal (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 3
Sepsis (Infections and infestations) | 1
Upper respiratory tract infection (Infections and infestations) | 1
Fall (Injury, poisoning and procedural complications) | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1
Anaplastic astrocytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Central nervous system lesion (Nervous system disorders) | 1
Cerebrovascular accident (Nervous system disorders) | 1
Hypoaesthesia (Nervous system disorders) | 1
Migraine (Nervous system disorders) | 1
Neurological symptom (Nervous system disorders) | 1
Sciatica (Nervous system disorders) | 1
Syncope (Nervous system disorders) | 1
Transient ischaemic attack (Nervous system disorders) | 1
Depression (Psychiatric disorders) | 1
Mental status changes (Psychiatric disorders) | 1
Renal failure acute (Renal and urinary disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Thyroidectomy (Surgical and medical procedures) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Nilotinib (N=128)
Anaemia (Blood and lymphatic system disorders) | 22
Leukopenia (Blood and lymphatic system disorders) | 7
Neutropenia (Blood and lymphatic system disorders) | 13
Thrombocytopenia (Blood and lymphatic system disorders) | 18
Palpitations (Cardiac disorders) | 8
Abdominal distension (Gastrointestinal disorders) | 7
Abdominal pain (Gastrointestinal disorders) | 24
Abdominal pain upper (Gastrointestinal disorders) | 12
Constipation (Gastrointestinal disorders) | 30
Diarrhoea (Gastrointestinal disorders) | 29
Dry mouth (Gastrointestinal disorders) | 13
Dyspepsia (Gastrointestinal disorders) | 10
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 7
Nausea (Gastrointestinal disorders) | 45
Vomiting (Gastrointestinal disorders) | 23
Asthenia (General disorders) | 7
Chest pain (General disorders) | 8
Fatigue (General disorders) | 58
Oedema peripheral (General disorders) | 9
Pyrexia (General disorders) | 8
Hyperbilirubinaemia (Hepatobiliary disorders) | 9
Bronchitis (Infections and infestations) | 8
Sinusitis (Infections and infestations) | 9
Upper respiratory tract infection (Infections and infestations) | 21
Urinary tract infection (Infections and infestations) | 8
Alanine aminotransferase increased (Investigations) | 19
Amylase increased (Investigations) | 10
Aspartate aminotransferase increased (Investigations) | 11
Blood bilirubin increased (Investigations) | 17
Lipase increased (Investigations) | 31
Weight increased (Investigations) | 8
White blood cell count decreased (Investigations) | 7
Decreased appetite (Metabolism and nutrition disorders) | 17
Hyperglycaemia (Metabolism and nutrition disorders) | 9
Hypomagnesaemia (Metabolism and nutrition disorders) | 8
Hypophosphataemia (Metabolism and nutrition disorders) | 8
Arthralgia (Musculoskeletal and connective tissue disorders) | 25
Back pain (Musculoskeletal and connective tissue disorders) | 10
Bone pain (Musculoskeletal and connective tissue disorders) | 9
Muscle spasms (Musculoskeletal and connective tissue disorders) | 22
Myalgia (Musculoskeletal and connective tissue disorders) | 23
Pain in extremity (Musculoskeletal and connective tissue disorders) | 12
Dizziness (Nervous system disorders) | 23
Headache (Nervous system disorders) | 31
Hypoaesthesia (Nervous system disorders) | 14
Paraesthesia (Nervous system disorders) | 9
Somnolence (Nervous system disorders) | 8
Anxiety (Psychiatric disorders) | 12
Depression (Psychiatric disorders) | 10
Insomnia (Psychiatric disorders) | 15
Cough (Respiratory, thoracic and mediastinal disorders) | 15
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 26
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 12
Alopecia (Skin and subcutaneous tissue disorders) | 22
Dry skin (Skin and subcutaneous tissue disorders) | 18
Night sweats (Skin and subcutaneous tissue disorders) | 9
Pruritus (Skin and subcutaneous tissue disorders) | 20
Rash (Skin and subcutaneous tissue disorders) | 48

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial or disclosure of trial results in their entirety.